CLINICAL TRIAL: NCT02965430
Title: PERFORMANCE STUDY OF THE AL-SENSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F-7-32.4-5.1
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2017-12

CONDITIONS: Amniotic Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL-SENSE diagnostic pantyliner (Experimental): AL-SENSE diagnostic pantyliner of amniotic fluid compared with standard clinical diagnosis methods.
  Interventions: Device: AL-SENSE

INTERVENTIONS:
Device: AL-SENSE — A diagnostic pantyliner for detection of amniotic fluid leaks compared with standard clinical diagnosis

SUMMARY:
This is an open-label, comparative, and prospective pivotal study to demonstrate that AL-SENSE can indicate whether wetness sensed by pregnant women may be caused by amniotic fluid leakage rather than by urinary incontinence.

Subjects arriving at the hospital will receive a single AL-SENSE to use until they notice any wetness.

The blinded physician will perform a diagnosis according to the standard diagnostic methods (clinical assessment). The standard diagnostic methods will include the following tests: (1) Pooling test, (2) Ferning test, (3) pH test by pH paper. A positive Pooling test or positive result in both the pH test and the Ferning test is defined as a positive clinical assessment.

DETAILED DESCRIPTION:
This is an open-label, comparative, and prospective pivotal study to demonstrate that AL-SENSE can indicate whether wetness sensed by pregnant women may be caused by amniotic fluid leakage rather than by urinary incontinence. Subjects arriving at the hospital and reporting unidentified wetness (undetermined whether this is amniotic fluid leakage or urinary incontinence) will receive a single AL-SENSE to use up to 12 hours or until they notice any wetness. The clinician will explain the proper use and handling of the AL-SENSE.

In each case, the blinded clinician will be required to read and record any occurrence of color change of the AL-SENSE 10 minutes after the AL-SENSE removal and to mark if it changes color to blue or to green on the designated form.

The blinded physician (other than the clinician who records the AL-SENSE results) will perform a diagnosis according to the standard diagnostic methods (clinical assessment). The standard diagnostic methods will include the following tests: (1) Pooling test, (2) Ferning test, (3) pH test by pH paper. A positive Pooling test or positive result in both the pH test and the Ferning test is defined as a positive clinical assessment.

In cases where the AL-SENSE shows positive results but the clinical assessment results are negative, reference laboratories, or any other standard procedure will check for the possibility of BV or Trichomonas in addition to the tests noted above.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or greater.
2. Subject minimum 16 weeks of pregnancy.
3. Who will sign the informed consent form.
4. Who arrive at the obstetric department reporting a feeling of vaginal wetness feeling (undetermined whether this is amniotic fluid leakage or urinary incontinence).

Exclusion Criteria:

1. Subject who has experienced intermittent vaginal bleeding between the 2nd and 3rd trimesters.
2. Subjects that have had sexual intercourse within the last 12 hours.
3. Subject is unable or unwilling to cooperate with study procedures.
4. Subject that has been diagnosed with Bacterial Vaginosis or Trichomonas infection within the last 3 days.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
color change of the pantyliner in comparison to standard clinical diagnosis | 10 min
  presence or absence of a blue or green stain on a yellow background as observed by the clinician yielded by the AL-SENSE in addition to the binary clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No